CLINICAL TRIAL: NCT03619746
Title: The Utility of a Point-of-Care Ultrasound Educational Initiative in Decreasing Unnecessary Antibiotic Use in Children With Local Reactions From Insect Bites
Brief Title: Point-of-Care Ultrasound Educational Initiative for Insect Bites
Acronym: USED4BUGBITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual. We were unable to enroll enough participants to have meaningful results.
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, James Meltzer, Associate Professor, Pediatrics, Jacobi Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-9176
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Cellulitis; Insect Bites; Insect Stings
Keywords: infection
MeSH Terms: conditions — Cellulitis; Insect Bites and Stings; Infections

STUDY DESIGN:
Intervention Model Description: Pre-Post Study Design with Non-Pharmacologic Intervention
  Patient in first arm of study will be treated by physicians who have not yet received educational training. Patients in the second arm of the study will be treated by physicians who went through the educational training.
Masking Description: All participants in the study (i.e., patients and physicians) will be aware of what arm of the study they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention (No Intervention): Current practice (unchanged). This arm of patients will cared for by physicians who have NOT received the POCUS Educational Intervention.
- Post-Intervention (Experimental): This arm of patients will cared for by physicians who have received the POCUS Educational Intervention.
  Interventions: Behavioral: POCUS Educational Intervention

INTERVENTIONS:
Behavioral: POCUS Educational Intervention — Midway through the study, all Pediatric Emergency Attendings and Fellows at Jacobi Medical Center will receive an educational session that describes how to properly perform a soft tissue examination using point-of-care ultrasound to differentiate between cellulitis and local allergic reaction.
  Arms: Post-Intervention

SUMMARY:
This pre-post study, designed to decrease unnecessary antibiotic prescribing, will use a prospective cohort of patients presenting to the Pediatric Emergency Department (PED). Patients with local skin findings that the clinician believes are primarily due to an insect bite or sting will be approached for the study.

The intervention will occur at the physician level. Midway through the study, physicians will receive an educational intervention describing how to differentiate cellulitis from allergic reaction using point-of-care bedside ultrasound.

The main outcome observed will be whether or not the patient receives a prescription for antibiotics at the index visit.

DETAILED DESCRIPTION:
Thousands of children each year develop soft tissue swelling after an insect bite or sting and present shortly after to emergency departments (ED) across the United States. These wounds are particularly pruritic and can become self-inoculated with skin flora resulting in cellulitis. Clinicians who suspect cellulitis will typically prescribe oral antibiotics to treat this condition. Cellulitis, however, can be confused with a local allergic reaction to the insect bite because the physical examination findings are nearly identical. As such, the reliability of clinical examination in the diagnosis of pediatric skin and soft tissue infections is poor. Consequently, many patients with local allergic reactions are treated unnecessarily with antibiotics.

Patients who take antibiotics may experience unintended and unpleasant side effects such as diarrhea and allergic reactions. Moreover, unnecessary antibiotic prescribing is an important factor in the development of antibiotic-resistant infections which are estimated to affect 2 million patients and result in 23 thousand deaths each year in the United States. The medical community has thus sought innovative approaches to reducing unnecessary antibiotic use.

The goal of this study is to reduce unnecessary antibiotic prescriptions for children with insect bites that are not infected. This quality improvement initiative will focus on children with insect bites presenting to the Pediatric Emergency Department at Jacobi Medical Center (Bronx, NY). The pre-intervention phase will consist of patients enrolled prior to the physicians receiving a Point-of-Care Ultrasound (POCUS) Educational Intervention. The post-intervention phase will consist of patients enrolled after the physicians have received a POCUS Educational Intervention. In both phases, the physician will be able to care for the patient however he or she believes is appropriate.

The POCUS Education Intervention will supplement the baseline knowledge of the Pediatric Emergency Medicine physician with regards to performing a soft-tissue examination using POCUS. A POCUS expert will train all clinicians how to properly perform a soft tissue examination using POCUS to differentiate between cellulitis and local reactions due to angioedema/allergic reaction. The education will include a formal lecture and practical clinical examination. The proportion of patients receiving antibiotics will be compared before and after the Educational Initiative had started. All patients will be contacted 3 to 5 days after their initial emergency department visit to determine if the patient's condition worsened, if the patient needed to return to a healthcare provider, and if the patient had taken any antibiotics.

ELIGIBILITY:
Inclusion Criteria:

- Erythema or swelling surrounding an insect bite or sting for greater than 12 hours

Exclusion Criteria:

* Patients with skin findings consistent with an abscess (ie. active drainage, fluctuance)
* Patients who are relatively immunocompromised (e.g., patients with AIDS, diabetes mellitus, cancer)
* Recent use of antibiotics within 1 week prior to symptoms
* Pregnant
* Altered mental status
* Unable to provide a phone number for follow-up

Ages: 3 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Antibiotic Prescription | index visit to the emergency department
  - whether or not the patient received a prescription for antibiotics prior to leaving the emergency department. This will be determined by review of the data collection instrument filled out by clinician at initial visit as well as review of the electronic medical record for that visit.

CONTACTS AND LOCATIONS:
Overall Officials: James A Meltzer, MD, MS, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Severino M, Bonadonna P, Passalacqua G. Large local reactions from stinging insects: from epidemiology to management. Curr Opin Allergy Clin Immunol. 2009 Aug;9(4):334-7. doi: 10.1097/ACI.0b013e32832d0668. PMID 19458526
- [Background] Blaabjerg S, Artzi DM, Aabenhus R. Probiotics for the Prevention of Antibiotic-Associated Diarrhea in Outpatients-A Systematic Review and Meta-Analysis. Antibiotics (Basel). 2017 Oct 12;6(4):21. doi: 10.3390/antibiotics6040021. PMID 29023420
- [Background] Solomon SL, Oliver KB. Antibiotic resistance threats in the United States: stepping back from the brink. Am Fam Physician. 2014 Jun 15;89(12):938-41. No abstract available. PMID 25162160
- [Background] Araujo da Silva AR, Albernaz de Almeida Dias DC, Marques AF, Biscaia di Biase C, Murni IK, Dramowski A, Sharland M, Huebner J, Zingg W. Role of antimicrobial stewardship programmes in children: a systematic review. J Hosp Infect. 2018 Jun;99(2):117-123. doi: 10.1016/j.jhin.2017.08.003. Epub 2017 Aug 12. PMID 28807835
- [Background] Sivitz AB, Lam SH, Ramirez-Schrempp D, Valente JH, Nagdev AD. Effect of bedside ultrasound on management of pediatric soft-tissue infection. J Emerg Med. 2010 Nov;39(5):637-43. doi: 10.1016/j.jemermed.2009.05.013. Epub 2009 Aug 8. PMID 19665335
- [Background] Tayal VS, Hasan N, Norton HJ, Tomaszewski CA. The effect of soft-tissue ultrasound on the management of cellulitis in the emergency department. Acad Emerg Med. 2006 Apr;13(4):384-8. doi: 10.1197/j.aem.2005.11.074. Epub 2006 Mar 10. PMID 16531602
- [Background] Subramaniam S, Bober J, Chao J, Zehtabchi S. Point-of-care Ultrasound for Diagnosis of Abscess in Skin and Soft Tissue Infections. Acad Emerg Med. 2016 Nov;23(11):1298-1306. doi: 10.1111/acem.13049. Epub 2016 Nov 1. PMID 27770490
- [Background] Tay ET, Tsung JW. Sonographic appearance of angioedema in local allergic reactions to insect bites and stings. J Ultrasound Med. 2014 Sep;33(9):1705-10. doi: 10.7863/ultra.33.9.1705. PMID 25154956
- [Background] American College of Emergency Physicians. Emergency ultrasound guidelines. Ann Emerg Med. 2009 Apr;53(4):550-70. doi: 10.1016/j.annemergmed.2008.12.013. No abstract available. PMID 19303521
- [Background] Marin JR, Bilker W, Lautenbach E, Alpern ER. Reliability of clinical examinations for pediatric skin and soft-tissue infections. Pediatrics. 2010 Nov;126(5):925-30. doi: 10.1542/peds.2010-1039. Epub 2010 Oct 25. PMID 20974788
- [Background] Marin JR, Dean AJ, Bilker WB, Panebianco NL, Brown NJ, Alpern ER. Emergency ultrasound-assisted examination of skin and soft tissue infections in the pediatric emergency department. Acad Emerg Med. 2013 Jun;20(6):545-53. doi: 10.1111/acem.12148. PMID 23758300
- [Background] Greenlund LJS, Merry SP, Thacher TD, Ward WJ. Primary Care Management of Skin Abscesses Guided by Ultrasound. Am J Med. 2017 May;130(5):e191-e193. doi: 10.1016/j.amjmed.2016.11.040. Epub 2016 Dec 22. PMID 28012823
- [Background] Adams CM, Neuman MI, Levy JA. Point-of-Care Ultrasonography for the Diagnosis of Pediatric Soft Tissue Infection. J Pediatr. 2016 Feb;169:122-7.e1. doi: 10.1016/j.jpeds.2015.10.026. Epub 2015 Nov 10. PMID 26563535
- [Background] Iverson K, Haritos D, Thomas R, Kannikeswaran N. The effect of bedside ultrasound on diagnosis and management of soft tissue infections in a pediatric ED. Am J Emerg Med. 2012 Oct;30(8):1347-51. doi: 10.1016/j.ajem.2011.09.020. Epub 2011 Nov 17. PMID 22100468
- [Background] Marin JR, Alpern ER, Panebianco NL, Dean AJ. Assessment of a training curriculum for emergency ultrasound for pediatric soft tissue infections. Acad Emerg Med. 2011 Feb;18(2):174-82. doi: 10.1111/j.1553-2712.2010.00990.x. PMID 21314777
- [Background] Vieira RL, Hsu D, Nagler J, Chen L, Gallagher R, Levy JA; American Academy of Pediatrics. Pediatric emergency medicine fellow training in ultrasound: consensus educational guidelines. Acad Emerg Med. 2013 Mar;20(3):300-6. doi: 10.1111/acem.12087. PMID 23517263
- [Background] Pallin DJ, Camargo CA Jr, Schuur JD. Skin infections and antibiotic stewardship: analysis of emergency department prescribing practices, 2007-2010. West J Emerg Med. 2014 May;15(3):282-9. doi: 10.5811/westjem.2013.8.18040. Epub 2014 Jan 6. PMID 24868305
- [Background] May L, Harter K, Yadav K, Strauss R, Abualenain J, Keim A, Schmitz G. Practice patterns and management strategies for purulent skin and soft-tissue infections in an urban academic ED. Am J Emerg Med. 2012 Feb;30(2):302-10. doi: 10.1016/j.ajem.2010.11.033. Epub 2011 Jan 28. PMID 21277138
- [Background] Haynes D, Lasarev M, Keller J. Systemic antibiotic use for nonbacterial dermatological conditions among referring providers. Int J Dermatol. 2018 May;57(5):566-571. doi: 10.1111/ijd.13962. Epub 2018 Mar 9. PMID 29521429
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059